CLINICAL TRIAL: NCT03325647
Title: TESTO: Testosterone Effects on Short-Term Outcomes in Infants With XXY
Acronym: TESTO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 17-1317; 5K23HD092588-02 (NIH)
Record Dates: First submitted 2017-10-16; First posted 2017-10-30 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-04

CONDITIONS: Klinefelter Syndrome
Keywords: body composition; klinefelter syndrome; XXY; sex chromosome variation; sex chromosome aneuploidy; testosterone
MeSH Terms: conditions — Klinefelter Syndrome

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Visit 1 Drug, Visit 2 Placebo (Experimental): Subjects in this group will be randomized to receive Testosterone Cypionate 200 Milligram/Milliliter Injectable Solution every 4 weeks x 3 doses, beginning at visit 1, and Placebo Injectable Saline beginning at visit 2.
  Interventions: Drug: Testosterone Cypionate 200 Milligram/Milliliter Injectable Solution; Drug: Placebo injectable saline
- Visit 1 Placebo, Visit 2 Drug (Experimental): Subjects in this group will be randomized to receive Placebo Injectable Saline beginning at visit 1, and Testosterone Cypionate 200 Milligram/Milliliter Injectable Solution every 4 weeks x 3 doses beginning at visit 2.
  Interventions: Drug: Testosterone Cypionate 200 Milligram/Milliliter Injectable Solution; Drug: Placebo injectable saline

INTERVENTIONS:
Drug: Testosterone Cypionate 200 Milligram/Milliliter Injectable Solution — Subjects in one arm will be randomized to receive testosterone cypionate 200 mg/ml intramuscularly every 4 weeks for a total of three doses after visit 1, and receive placebo injectable saline for the same duration starting at visit 2. Subjects in the other arm will be randomized to receive placebo injectable saline every 4 weeks for a total of 3 doses after visit 1, and testosterone cypionate 200 mg/ml intramuscularly for the same duration starting at visit 2.
Drug: Placebo injectable saline — Subjects in one arm will be randomized to receive testosterone cypionate 200 mg/ml intramuscularly every 4 weeks for a total of three doses after visit 1, and receive placebo injectable saline for the same duration starting at visit 2. Subjects in the other arm will be randomized to receive placebo injectable saline every 4 weeks for a total of 3 doses after visit 1, and testosterone cypionate 200 mg/ml intramuscularly for the same duration starting at visit 2.

SUMMARY:
This research study in infant males with Klinefelter syndrome (47,XXY) will learn more about the effect of testosterone on early health and development. The study is a total of three visits over 6 months with assessments of motor skills, body composition (muscle and fat), and hormone levels. This is a randomized, placebo-controlled study but all infants will receive testosterone treatment during the study period. The investigators will learn how testosterone treatment in infancy effects short term outcome measures on health and development.

DETAILED DESCRIPTION:
XXY (also known as Klinefelter syndrome) is the most common chromosomal abnormality in males, affecting 1/600 boys. The extra X chromosome leads to insufficient development of the testicles and subsequent testosterone deficiency. Males with XXY also have a high risk for developmental delays, learning disabilities, and cardiovascular disease. An essential question is how much of this risk is because of testosterone deficiency and could therefore be reduced by testosterone supplementation, particularly during critical periods of development.

In typical male development, there is a surge of testosterone in the first few months of life, commonly known as the "mini-puberty period of infancy." This testosterone surge may be critical for neurodevelopmental and cardiometabolic programming throughout life. Recently there has been increased off-label use of testosterone in infants with XXY, however neither the short or long term safety or efficacy have been evaluated. This study aims to quantify the short term effects of testosterone treatment in infants with XXY on neurodevelopment, growth, body composition, testicular function, and safety parameters. This is a double blind randomized placebo controlled trial of testosterone injections 25 mg every 4 weeks for 3 doses in boys with XXY enrolled between 1 and 3 months of age. Outcomes including body fat percentage, scaled motor developmental scores, growth velocity, testicular hormone concentrations, specific metabolites, and safety parameters will be assessed 12 weeks into the study. The groups will then cross-over (all subjects will receive testosterone during the study period) and the outcomes will be reassessed 24 weeks into the study. The secondary questions the investigators will answer with this cross-over is 1) whether benefits in the treatment group at 12 weeks are sustained at 24 weeks, and 2) whether the same benefits are seen if treated after the mini-puberty period.

ELIGIBILITY:
Inclusion Criteria:

* Male infants with 47,XXY karyotype identified prenatally who are 4-12 weeks old (31 to 90 days of age). 47,XXY must be from a diagnostic test such as Chorionic Villus Sampling (CVS), amniocentesis, or post-natal blood/tissue. Non-invasive prenatal screening results alone will not be accepted.

Exclusion Criteria:

* >20 percent mosaicism for a normal cell line
* Gestational age at birth <36 weeks
* Birth weight <2.5th percentile or >97.5 percentile for age (small or large for gestational age)
* History of thrombosis in self or a first degree relative
* Exposure to androgen therapy outside the study protocol
* Use of medications known to affect body composition, such as growth hormone or insulin
* Known allergy to the testosterone cypionate solution components including benzyl benzoate, benzyl alcohol, or cottonseed oil

Ages: 31 Days to 90 Days | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Change in Body Fat Percentage | Baseline and 3 months
  Body fat percentage will be measured using air displacement plethysmography (PEA POD) at the beginning and end of the study period
Change in Composite Motor Score on Alberta Infant Motor Scale | 3 months
  Motor development will be assessed using the standardized Alberta Infant Motor Scale
Change in C14:1 Long Chain Acylcarnitines (LCAC) through targeted metabolomics | Baseline and 3 months
  Plasma will be processed and stored until batch analysis using electrospray tandem mass spectroscopy per standard protocols to quantify acylcarnitines (short, medium, and long-chain) and Branched-Chain Amino Acids (BCAA--leucine/isoleucine and valine) at baseline and 12 weeks.

SECONDARY OUTCOMES:
Change in height | 6 months
  Physical exam measurements will be measured by a physician at each visit
Change in weight | 6 months
  Physical exam measurements will be measured by a physician at each visit
Change in weight-for-length | 6 months
  Physical exam measurements will be measured by a physician at each visit
Change in waist circumference | 6 months
  Physical exam measurements will be measured by a physician at each visit
Change in serum leptin | 6 months
  Serum will be collected and measured at each study visit.
Change in lipids | 6 months
  Serum will be collected and measured at each study visit.
Change in insulin | 6 months
  Serum will be collected and measured at each study visit.
Change in serum Luteinizing Hormone (LH) | 6 months
  Serum will be collected at each study visit. Ultrasensitive LH will be measured.
Change in serum Follicle Stimulating Hormone (FSH) | 6 months
  Serum will be collected at each study visit. Follicle Stimulating Hormone (FSH) will be measured.
Change in Inhibin B (INHB) | 6 months
  Inhibin B levels will be measured.
Change in Anti-Mullerian Hormone (AMH) | 6 months
  Serum will be collected at each study visit. AMH levels will be measured.
Change in Total Testosterone (Total T) | 6 months
  Serum will be collected at each study visit. Total testosterone by mass spectroscopy will be measured.
Change in Gross Motor Scores on the Peabody Developmental Motor Scales 2 | 6 months
  Gross motor development will be assessed using the standardized Peabody Developmental Motor Scales 2. The Peabody Developmental Motor Scales 2 measures gross motor development using the subscale of the Gross Motor Quotient, which measures the ability to utilize the large muscle systems. High scores on this composite are made by children with well-developed gross motor abilities.
Change in Gross Motor Scores on the Alberta Infant Motor Scales | 6 months
  Gross motor development will be assessed using the standardized Alberta Infant Motor Scales (AIMS). The Alberta Infant Motor Scales is a performance-based and norm-referenced measure of infant gross motor maturation from birth to 18 months. The AIMS total score is calculated by summing the scores for the 58 items, with the score ranging between 0 and 58. Higher scores indicate more mature motor development. The infant's score can then be converted to a percentile and compared with age-equivalent peers from the normative sample.
Change in Fine Motor Scores | 6 months
  Fine motor development will be assessed using the standardized Peabody Developmental Motor Scales 2. The Peabody Developmental Motor Scales 2 measures fine motor development using subscale of the Fine Motor Quotient, which measures a child's ability to use his or her hands and arms to grasp objects, stack blocks, draw figures, and manipulate objects. High scores on this composite are made by children with well-developed fine motor abilities.
Change in Cognitive and Language Composite Scores on the Bayley III | 6 months
  Cognition and language will be assessed by a trained administrator of developmental tests using the standardized Bayley Scales of Infant and Toddler Development III: cognitive and language domains. In each subscale, age-standardized scores are calculated using test norms. Developmental delay is determined by calculating how many standard deviations a child scores from the mean in that subscale. Typically, the more standard deviations below the mean, the more severe the delay.
Change in Adaptive Functioning | 6 months
  Adaptive Functioning will be assessed using the Adaptive Behavior Assessment System, 3rd edition, completed by the parent about their child.
Change in Number and Type of Adverse Events | 6 months
  Adverse events will be measured by verbal questionnaire and parent-report, to determine safety.
Change in Serum BCAA, other LCAC | 6 months
  BCAA and other LCAC will be measured through targeted metabolomics from serum collection at each visit.
Change in Pathway analysis | 3 months
  Serum Pathways will be measured through untargeted/unbiased metabolomics

CONTACTS AND LOCATIONS:
Overall Officials: Shanlee M Davis, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT03325647/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT03325647/ICF_001.pdf